CLINICAL TRIAL: NCT05750979
Title: Quantifying Disease Progression in Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation (LBSL)
Brief Title: Quantifying Disease Progression in LBSL
Acronym: LBSL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M. Engelen (Other)
Responsible Party: Sponsor-Investigator, M. Engelen, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: LBSL
Record Dates: First submitted 2023-02-18; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: LBSL; Leukoencephalopathies
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Leukocytes PAXGene for RNA storage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leukoencephalopathy with brain stem involvement and lactate elevation (LBSL) is a genetic disorder caused by biallelic mutations in the DARS2 gene that encodes mitochondrial aspartyl tRNA synthase.(1, 2) It is characterized by typical abnormalities on MRI of the brain and spinal cord.(3) Clinically, the disorder is heterogeneous and can present in the neonatal period, later in childhood or even in adults.(3) In general it can be stated that the earlier presentations are characterized by rapid progression leading to severe disability and death. Presentation at a later age is typically characterized by a more benign disease course, although considerable disability is common. Clinically, the disease presents as a slowly progressive myelopathy with mainly involvement of the corticospinal tracts and the dorsal columns. Although the natural history has been studied in large cohorts, the rate of progression has not been systematically studied with clinimetric outcome scales or potential surrogate outcomes for spinal cord disease.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age > 16 years
* Definite diagnosis of LBSL confirmed by DARS2 mutation analysis.
* Able to understand Dutch or English and provide informed consent.
* No contra-indications for MRI of brain and spinal cord.

Subjects eligible to participate as healthy controls must meet all of the following criteria:

* Willing to visit the hospital
* 16 years or older
* Provision of written informed consent to participate in the study obtained from the participant

For the MRI controls:

- No contra-indications for MRI of the brain and spinal cord

A potential subject (patient or healthy control) who meets any of the following criteria will be excluded from participation in this study:

* Unable to visit the hospital for the follow-up visits
* Co-existing neurological disease that can cause pyramidal tract signs making interpretation of acquired data difficult (for instance, multiple sclerosis, stroke, etc)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: LBSL patients and healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is disease progression on all parameters | 5 years
  disease progression

CONTACTS AND LOCATIONS:
Overall Officials: M. Engelen, Dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided